CLINICAL TRIAL: NCT04234386
Title: GCC 1926- Phase Ib Dose Escalation of Single-Fraction Preoperative Stereotactic Partial-Breast Irradiation for Early-Stage Breast Cancer
Brief Title: GammaPod Dose Escalation Radiation for Early Stage Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HP-00084710
Record Dates: First submitted 2020-01-08; First posted 2020-01-21 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Dose Level 1: 21 Gy (Active Comparator): Participants will receive radiation therapy to the partial breast using the GammaPod technology before a lumpectomy.
  Interventions: Radiation: GammaPod Radiation
- Dose Level 2: 24 Gy (Active Comparator): Participants will receive radiation therapy to the partial breast using the GammaPod technology before a lumpectomy.
  Interventions: Radiation: GammaPod Radiation
- Dose Level 3: 27 Gy (Active Comparator): Participants will receive radiation therapy to the partial breast using the GammaPod technology before a lumpectomy.
  Interventions: Radiation: GammaPod Radiation
- Dose Level 4: 30 Gy (Active Comparator): Participants will receive radiation therapy to the partial breast using the GammaPod technology before a lumpectomy.
  Interventions: Radiation: GammaPod Radiation

INTERVENTIONS:
Radiation: GammaPod Radiation — The basic design is a dose-escalation phase Ib study with 4 predefined dose levels. With this study treatment, participants will receive the dose level assigned treatment of radiation therapy before the lumpectomy surgery.

SUMMARY:
The GammaPod machine was made by Xcision Medical Systems and is already FDA cleared to deliver focused radiation within the breast. Unlike current radiation machines, the GammaPod was designed specifically for treating breast cancer. The GammaPod can pinpoint radiation to the tumor bed in the breast which lowers the amount of radiation to nearby tissues. The machine uses a breast cup system to hold the breast in place for the treatment. This breast cup system was tested at MSGCCC (Marlene Stewart Greenebaum Comprehensive Cancer Center). Patients reported this system was more comfortable than an MRI or mammogram. The cup system was able to securely position the breast for treatment in the correct location.

Receiving radiation before surgery is not a new concept in cancer management. Preoperative radiation has proven to result in improved disease free survival in certain types of cancer.

With this study treatment, the participants will receive a dose of breast radiation therapy before the lumpectomy surgery. The lumpectomy surgery is where they remove the participant's tumor.

The purpose of this research study is to determine a safe and effective dose of pre-operative radiation to treat early stage breast cancer. The pre-operative radiation is delivered using the FDA approved, GammaPod machine. The study will also determine the cosmesis of pre-operative radiation at different doses. Cosmesis is another word for looking at skin changes. The research team will use questionnaires for patient and physicians to assess adverse cosmesis changes as accurately as possible. In addition, the investigators are going to assess radiation related changes using photo software analysis tools and patients quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients must sign consent for study participation.
* Patients must be female with a diagnosis of invasive ductal carcinoma. Lobular histologies will not be included, because of difficulty in defining the extent of disease with imaging.
* Patients must be deemed appropriate candidates for breast-conserving therapy (i.e., not pregnant, never had RT to the treated breast, breast size would allow adequate cosmesis after volume loss from partial mastectomy).
* Tumor must not involve the overlying skin or underlying chest wall, based on imaging evaluation and/or clinical exam.
* Greatest tumor dimension is <3 cm based on US. MR imaging measurements can be included only if performed BEFORE the biopsy (postbiopsy measurements can be larger as a result of hematoma formation or increased edema).
* Tumor must be unifocal.
* Patients must be > 45 years old.
* The tumor must be visible on a CT scan.
* Patients must undergo MR imaging for work-up to aid in tumor delineation and to rule out additional foci of disease. If additional foci of disease are found to be present, then these must be biopsied with negative results to proceed with treatment.
* The tumor must be clinically and radiographically N0 (node negative). If a suspicious node is visualized, it must be biopsied with negative results.
* Patients must be estrogen-receptor positive.
* Patients must be HER2neu negative.
* Patients must weigh <150 kg (330 lb), which is the limit of the imaging loader.
* Patients must be <6'6" in height, again because of instrumentation limitations.
* Patients must be able to lie prone for treatment.
* Patients must have no lymphovascular invasion on biopsy.
* Patients may be taking hormonal therapy prior to initiation of treatment. This will be documented.

Exclusion Criteria:

* Multicentric disease.
* Prior RT to the involved breast.
* Inability to fit into the immobilization breast cup because of breast size or other anatomic reasons.
* Inability to obtain an adequate seal when using the immobilization breast cup.
* Male sex.
* Breast implants.
* Patient cannot comfortably lie in the prone position (i.e., physical disability).
* Patients who are planned to be treated surgically with a mastectomy.
* Tumor <5 mm from the skin surface or chest wall on clinical exam and/or radiographic imaging.
* Tumor size >3 cm.
* Patients with psychiatric or addictive disorders that would preclude obtaining informed consent or study completion.
* Patients who are pregnant or lactating (because of potential RT exposure to the fetus and unknown effects of RT in lactating women).
* Patient unable to undergo MR imaging (e.g., because of known contrast reaction or concerns about contrast and existing health status).
* Lymphovascular invasion on original biopsy.
* Tumor histologies other than invasive ductal carcinoma (including invasive lobular carcinoma).
* ER-negative tumors.
* HER2neu-positive tumors.
* Pure ductal carcinoma in situ (no invasive component).
* Weight >330 lb
* Prior ipsilateral breast cancer.
* Diffuse calcifications on mammogram (BIRADS 3, 4, 5).

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Establish the single-fraction radiation dose (MTD) | 5 years
  To establish the single-fraction radiation dose (MTD) delivered with the GammaPod that causes an incidence of dose-limiting toxicities (DLTs) that is statistically significantly 10% or lower.
Incidence of Dose-Limiting Toxicities (DLTs) | 5 years
  The primary endpoint is DLTs defined as one or more instances of:
  * Surgical infection: Defined as redness that resolves on antibiotics (sometimes the surgical site may look red as a result of natural healing processes and does not resolve with antibiotics) with or without fever and/or elevated white blood cell count. The risk of infection for this surgical procedure (lumpectomy ± SLN biopsy) is <5%.
  * Nonhealing surgical incision (>30 days). The risk is <5%.
  * Reoperation secondary to infection/wound healing problem. Risk is <5%.

SECONDARY OUTCOMES:
Establish a Comprehensive Safety Profile of single-fraction PBI delivered with the GammaPod | 5 years
  To establish the comprehensive safety profile of single-fraction PBI delivered with the GammaPod. The following secondary toxicity and quality-of-life endpoints will be collected and reported:
  * Acute toxicity (NCI-CTCAE v 5), including skin toxicity and fatigue.
  * Late toxicity (NCI-CTCAE v 5), including rates of fat necrosis.
Establish a Comprehensive Safety Profile of single-fraction PBI delivered with the GammaPod | 5 years
  To establish the comprehensive safety profile of single-fraction PBI delivered with the GammaPod. The following secondary toxicity and quality-of-life endpoints will be collected and reported:
  -Rates of surgical morbidity (defined below), including seroma formation. Seroma will be defined as any palpable seroma on follow-up exam. If seroma results in pain/discomfort and/or requires drainage this should be noted as a 'symptomatic' seroma. Seroma formation is normal following lumpectomy surgery but is asymptomatic in the majority of cases.
Establish a Comprehensive Safety Profile of single-fraction PBI delivered with the GammaPod | 5 years
  To establish the comprehensive safety profile of single-fraction PBI delivered with the GammaPod. The following secondary toxicity and quality-of-life endpoints will be collected and reported:
  -Patient and physician-assessed cosmesis after radiotherapy and surgery via questionnaire.
Establish a Comprehensive Safety Profile of single-fraction PBI delivered with the GammaPod | 5 years
  To establish the comprehensive safety profile of single-fraction PBI delivered with the GammaPod. The following secondary toxicity and quality-of-life endpoints will be collected and reported:
  - Patient Quality of Life Assessments [EORTC QLQ-C30- scale goes from 1/not at all to 4/very much. There is additionally a rate of overall health and quality of life that is a scale from 1 to 7.]
Rate of pathologic complete response (pCR) | 5 years
  To establish the rate of pathologic complete response (pCR) as a function of dose. pCR will be scored by pathology review of H&E slides.
Rate of ipsilateral local tumor recurrence | 5 years
  Report ipsilateral local tumor recurrence using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Nichols, MD, Principal Investigator — University of Maryland, Baltimore
Locations (4):
- United States (4):
  - UMMC, Baltimore, Maryland
  - Upper Chesapeake Health, Bel Air, Maryland
  - Central Maryland Oncology Center, Columbia, Maryland
  - Baltimore Washington Medical Center, Glen Burnie, Maryland

IPD SHARING:
Plan to Share IPD: No